CLINICAL TRIAL: NCT00619827
Title: A Randomised, Double-blind, in Parallel Groups Placebo-controlled, Mono-centre, Phase I Study to Assess After Allergen Challenge in an Allergen Exposition Chamber the Effect and Its Time Course of Sublingual Immunotherapy (SLIT) Administered as 300IR Allergen-based Tablets Once Daily to Adults Suffering From Grass Pollen Rhinoconjunctivitis
Brief Title: Efficacy and Safety of Sublingual Tablets of Grass Pollen Allergen Extract
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stallergenes Greer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VO56.07 A
Record Dates: First submitted 2008-02-08; First posted 2008-02-21 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-04

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Sublingual immunotherapy; Rhinitis; Conjunctivitis; Allergen challenge; Allergen exposition chamber; Grass pollen tablet; Allergic rhinoconjunctivitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis; Conjunctivitis | interventions — Sublingual Immunotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 300 IR (Experimental): 300 IR grass pollen allergen extract tablet
  Interventions: Drug: 300 IR grass pollen allergen extract tablet
- Placebo (Placebo Comparator): Placebo tablet
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: 300 IR grass pollen allergen extract tablet — 300 IR grass pollen allergen extract tablet once daily during four months
  Other Names: Sublingual immunotherapy tablet
  Arms: 300 IR
Drug: Placebo tablet — Placebo tablet once daily during four months
  Other Names: Sublingual placebo tablet
  Arms: Placebo

SUMMARY:
The objective of this study is to assess the effect of grass pollen extract SLIT tablets on the Rhinoconjunctivitis Total Symptom Score (RTSS) of the six rhinoconjunctivitis symptoms in response to grass pollen challenge after one week, one, two and four months of treatment in patients suffering from Seasonal Allergic Rhinoconjunctivitis (SAR) due to grass pollen.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether SLIT tablets are effective on symptoms of allergic rhinitis compared to placebo in patients suffering from allergic rhinitis to grass pollen when exposed in an allergen chamber and also to determine the onset of action of SLIT tablets on allergic rhinitis symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients 18-50 years old
* grass pollen rhinoconjunctivitis of at least 2 years.
* positive specific skin prick test and a specific IgE dosage level of at least 0.70 kU/L at screening.
* written consent
* a positive response to the baseline challenge test (RTSS reaches 7 at one time-point at least during baseline challenge)

Exclusion Criteria:

* Allergic rhino-conjunctivitis due to a co-sensitisation, likely to significantly change the symptoms of the subject throughout the study
* Asthma requiring treatment other than short-acting beta-2 inhaled agonists.
* Desensitisation treatment for grass pollen in the previous five years and current immunotherapy with another allergen.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2007-09; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Friedrich HORAK, Pr. MD, Principal Investigator — Allergy Center Vienna West, VIENNA, AUSTRIA
Locations (1):
- Allergy Center Vienna West, Vienna Challenge Chamber -, Vienna, Austria

REFERENCES:
- [Result] Horak F, Zieglmayer P, Zieglmayer R, Lemell P, Devillier P, Montagut A, Melac M, Galvain S, Jean-Alphonse S, Van Overtvelt L, Moingeon P, Le Gall M. Early onset of action of a 5-grass-pollen 300-IR sublingual immunotherapy tablet evaluated in an allergen challenge chamber. J Allergy Clin Immunol. 2009 Sep;124(3):471-7, 477.e1. doi: 10.1016/j.jaci.2009.06.006. Epub 2009 Aug 3. PMID 19647862
- [Derived] Baron-Bodo V, Horiot S, Lautrette A, Chabre H, Drucbert AS, Danze PM, Senechal H, Peltre G, Galvain S, Zeldin RK, Horak F, Moingeon P. Heterogeneity of antibody responses among clinical responders during grass pollen sublingual immunotherapy. Clin Exp Allergy. 2013 Dec;43(12):1362-73. doi: 10.1111/cea.12187. PMID 24261946
- [Derived] Bonvalet M, Moussu H, Wambre E, Ricarte C, Horiot S, Rimaniol AC, Kwok WW, Horak F, de Beaumont O, Baron-Bodo V, Moingeon P. Allergen-specific CD4+ T cell responses in peripheral blood do not predict the early onset of clinical efficacy during grass pollen sublingual immunotherapy. Clin Exp Allergy. 2012 Dec;42(12):1745-55. doi: 10.1111/cea.12015. PMID 23181790

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient First Visit 17 SEP 2007, Last Patient Last Visit 10 MAR 2008
Period: Overall Study
Arm/Group | 300 IR | Placebo
Started | 45 | 44
Completed | 42 | 40
Not Completed | 3 | 4
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) population included all randomised subjects who received at least one dose of the investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | 300 IR | Placebo | Total
Number analyzed (Participants) | 45 | 44 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.46 (6.577) | 27.12 (5.807) | 27.29 (6.175)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 28 | 52
  Male | 21 | 16 | 37

OUTCOME MEASURES:

1. Primary Outcome: Average of Rhinoconjunctivitis Total Symptom Score (ARTSS) ]0-4] Hours
Description: The primary efficacy variable was the Average of Rhinoconjunctivitis Total Symptom Score (ARTSS) during the four-hour (]0-4] hours) grass pollen allergen challenge at end point (after four months of treatment) of the 6 rhinoconjunctivitis symptoms (sneezing, rhinorrhea, nasal pruritus, nasal congestion, ocular pruritus and watery eyes). The severity of each symptom was evaluated by the subject, before allergen exposure and every 15 minutes during allergen challenge on a scale of 0 to 3; 0: no symptoms, 1: mild symptoms, 2: moderate symptoms, 3: severe symptoms, total score range was 0 to 18. The ARTSS ]0-4] hours was calculated as the mean of the RTSSs at each timepoint during the allergen challenge (i.e., 16 timepoints from 15 minutes to 4 hours) after 4 months of treatment (endpoint). The lower the score, the better the outcome.
Time Frame: 4 months
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: Units on a scale (range: 0 to 18)
Arm/Group | 300 IR | Placebo
Number analyzed (Participants) | 45 | 44
Units on a scale (range: 0 to 18) | 4.88 (0.363) | 6.84 (0.367)
Statistical Analysis 1: Comparison: 300 IR vs Placebo; Test type: Superiority or Other; p = 0.0003, ANCOVA; Mean Difference (Final Values) = -1.97, 95% CI 2-sided [-2.99 to -0.94]

ADVERSE EVENTS:
Time Frame: 4 months.
Description: A Treatment Emergent Adverse Event (TEAE) is defined as any adverse event that started on or after the first intake of the investigational product.
  Note: Serious Adverse Events and Other Adverse Events are described in the Results Publication.
Arm/Group | 300 IR | Placebo
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/44
Other Adverse Events (participants affected / at risk) | 24/45 | 9/44
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 300 IR (N=45) | Placebo (N=44)
Ear pruritus (Ear and labyrinth disorders) | 3 | 0
Oral pruritus (Gastrointestinal disorders) | 16 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 16 | 0
Headache (Nervous system disorders) | 8 | 8
Nasopharyngitis (Infections and infestations) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No